CLINICAL TRIAL: NCT04428502
Title: Correlation of Anti-CCP With Disease Activity and Its Impact on Biological Response in PsA in Iraqi Patients
Brief Title: Study To Evaluate The Impact Of Anti-Cyclic Citrullinated Peptide(Anti-CCP) For Management With Enbrel In Patients With Psoriatic Arthritis(PsA)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801418
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with psoriatic arthritis: Iraqi patients diagnosed with psoriatic arthritis that receive Enbrel as treatment for disease
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — As provided in real world practice

SUMMARY:
This study is to evaluate the local data in Iraqi patients with psoriatic arthritis on Enbrel treatment with positive Anti-Cyclic Citrullinated Peptide using data from the Rheumatologist in Baghdad Teaching Hospital registry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PsA patients.
* ≥18 years of age
* Have not received previous biological treatment

Exclusion Criteria:

* Previous use of other biological treatments.
* Etanercept use for less than 1 year duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from the local Rheumatology Center of Baghdad Teaching Hospital registry
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801418

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data of Iraq's participants, 1) who aged greater than or equal to (>=) 18 years, 2) who met American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 criteria for psoriatic arthritis (PsA), and 3) who received etanercept for at least for 1 year from May 2012 until August 2019 in the Baghdad teaching hospital (rheumatology center) were collected. Data collected were assessed in approximately 1.8 months of this retrospective observational study.
Groups:
- Etanercept: Participants received etanercept to treat PsA at least for 1 year from May 2012 until August 2019 under standard clinical practice. Data of these participants was studied for approximately 1.8 months.
Period: Overall Study
Arm/Group | Etanercept
Started | 127
Completed | 113
Not Completed | 14
Not completed — Did not meet entrance criteria | 14

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants who were included in this study.
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity in Psoriatic Arthritis (DAPSA) Score at Month 1
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), C-reactive protein (CRP) level (milligram per deciliter [mg/dL]), participant assessment of pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and participant's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0= excellent and 10= poor). A higher DAPSA score indicated more active disease activity. The assessment did not have a score range with an upper or lower bound. The outcome measure compared response between anti-cyclic citrullinated peptide positive and negative participants.
Time Frame: Baseline, Month 1
Population: Data was not evaluated and reported for this outcome measure since CRP variable to calculate DAPSA was not collected from the participants.
Groups:
- Etanercept: ACCP Positive: Participants received etanercept to treat PsA at least for 1 year from May 2012 until August 2019 under standard clinical practice and had positive ACCP status.
- Etanercept: ACCP Negative: Participants received etanercept to treat PsA at least for 1 year from May 2012 until August 2019 under standard clinical practice and had negative ACCP status.
Arm/Group | Etanercept: ACCP Positive | Etanercept: ACCP Negative
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in Disease Activity in Psoriatic Arthritis (DAPSA) Score at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: as for outcome 1
Arm/Group | Etanercept: ACCP Positive | Etanercept: ACCP Negative
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Disease Activity Score 28 Erythrocyte Sedimentation Rate (DAS28 ESR) at Month 1, 6 and 12
Description: DAS28 ESR was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, ESR (millimeters per hour [mm/hour]) and participant's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS 28 ESR =0.56*sqrt (PJC28) + 0.28*sqrt (SJC28) + 0.70*In (ESR) + 0.014*PtGA; ln = natural logarithm, sqrt = square root of. DAS28 ESR less than equal to (<=) 3.2 = low disease activity, DAS28 ESR greater than (>) 3.2 to 5.1 = moderate to high disease activity. The outcome measure compared response between anti-cyclic citrullinated peptide positive and negative participants.
Time Frame: Month 1, 6 and 12
Population: Analysis was performed on all participants who were included in this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: ACCP Positive | Etanercept: ACCP Negative
Number analyzed (Participants) | 20 | 107
units on a scale
  Month 1 | 4.2 (0.77) | 4.1 (0.8)
  Month 6 | 4.06 (0.93) | 3.35 (1.08)
  Month 12 | 3.34 (1.1) | 2.66 (0.91)
Statistical Analysis 1: Comparison: Etanercept: ACCP Positive vs Etanercept: ACCP Negative; At Month 1: P-value <0.05 was considered statistically significant, without multiplicity adjustment; Test type: Equivalence — Hypothesis tested was to evaluate that there is no difference in response between ACCP positive and ACCP negative PsA participants who were treated with etanercept; p = 0.6, Student's t-test
Statistical Analysis 2: Comparison: Etanercept: ACCP Positive vs Etanercept: ACCP Negative; At Month 6: P-value <0.05 was considered statistically significant, without multiplicity adjustment; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.007, Student's t-test
Statistical Analysis 3: Comparison: Etanercept: ACCP Positive vs Etanercept: ACCP Negative; At Month 12: P-value <0.05 was considered statistically significant, without multiplicity adjustment; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.004, Student's t-test

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) was not met, hence adverse events were not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04428502/Prot_SAP_000.pdf